CLINICAL TRIAL: NCT00764491
Title: OptiMesh® for Lumbar Interbody Fusion Trial (OLIF)
Acronym: OLIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spineology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G030106
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
Keywords: Degenerative Disc Disease; DDD; Lumbar DDD; Disc degeneration; Interbody Fusion; Lumbar Interbody Fusion; IBF
MeSH Terms: conditions — Intervertebral Disc Degeneration; Dowling-Degos Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Optimesh 1500S (Experimental): OptiMesh 1500S, filled with a mixture of demineralized bone matrix (DBM) and cortico-cancellous bone, placed into the interbody space from the posterior approach and supplemental pedicle screws.
  Interventions: Device: OptiMesh 1500S
- Structural Allograft Spacer (Active Comparator): Structural Allograft Spacer with pedicle screws.
  Interventions: Device: Structural Allograft Spacer

INTERVENTIONS:
Device: Structural Allograft Spacer — Following disc space preparation the spacer is placed in accordance with cleared labeling and supplemental instrumentation is provided as an adjunct to fixation.
  Other Names: Allograft bone spacer
  Arms: Structural Allograft Spacer
Device: OptiMesh 1500S — Following disc space preparation the OptiMesh is deployed and filled in accordance with study surgical technique and supplemental instrumentation is provided as an adjunct to fixation.
  Other Names: OptiMesh; OLIF
  Arms: Optimesh 1500S

SUMMARY:
The purpose of this study was to collect data to demonstrate the safety and effectiveness of the OptiMesh 1500S to contain and reinforce bone graft materials in patients with Degenerative Disc Disease (DDD) whose condition requires an interbody spinal fusion procedure combined with posterior fixation.

DETAILED DESCRIPTION:
Seventy-six thousand posterior interbody fusions are performed annually in the U.S., and it has been estimated that at least 50% of those cases include supplemental posterior instrumentation. For interbody fusion with posterior fixation, spine surgeons currently place structural intervertebral spacers into the interbody space. These spacers may be pre-shaped devices constructed of allograft (cortical bone dowels or femoral rings) or non-metallic, radiolucent materials, or metallic cage devices. Autogenous bone graft and blood components (marrow, blood) are often added.

Use of morselized bone graft in orthopedic procedures is desirable because it is more rapidly incorporated during the course of bone healing. If the morselized graft pack can be effectively contained in the interbody space, the graft material can function as a structural spacer to provide anterior column support. Contained graft material can be tightly packed within the mesh to increase the graft's compressive strength. Unlike pre-shaped cortical grafts, the morselized pack conforms intimately to the host bone at the surgical site, ensuring good vascularization potential and reducing the osteoblast jumping distance for osteogenesis. In addition, the solidly packed graft retains intra-pack porosity, ensuring an osteoconductive scaffold to facilitate vascular and bony ingrowth.

It would be desirable to minimize autograft use because of associated post-op pain, to optimize contact between allograft and host bone, and to permit the surgeon to place or construct an effective structural intervertebral spacer with only minimal neural retraction required.

OptiMesh 1500S is intended to be used to contain the bone graft placed by spine surgeons into the interbody space to achieve spinal intervertebral body fusion. OptiMesh 1500S enables the use of morselized bone graft materials in spine fusion procedures instead of solid allograft materials, such as cortical bone dowels or femoral rings, or rigid synthetic materials.

In addition, the OptiMesh instrument system allows the surgeon to perform an interbody fusion through a small portal and to complete the entire fusion procedure from a posterior approach instead of a 360 degree anterior/ posterior procedure, which is often the case with the use of cages. The minimal access portal utilized for OptiMesh filling allows the device to be placed via a unilateral transforaminal or translaminar approach, versus the often-used bilateral approach required for many cages and cortical spacers. This flexibility permits the surgeon to adapt the surgical approach to the local anatomy of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature and be at least 18 years of age
* Have degenerative disc disease (DDD) requiring one level fusion between L2 and S1, with DDD confirmed by subject history, physical exam, and radiographic studies with one or more of the following factors:

  1. instability as defined by >3 mm translation or ≥5º rotation of flexion/ extension;
  2. osteophyte formation of facet joints or vertebral endplates;
  3. decreased disc height, on average 2 mm, but dependent on spinal level;
  4. scarring/thickening of the ligamentum flavum, annulus fibrosis, or facet joint capsule;
  5. herniated nucleus pulposus;
  6. facet joint degeneration/changes; and/or
  7. vacuum phenomenon;
* Based on the VAS, subjects report pre-operative low back pain (>4 of 10) with duration of pain six-months or longer despite non-surgical treatment;
* Capable of understanding and signing the consent form; and
* Willing and able to comply with follow-up requirements

Exclusion Criteria:

* A previous interbody fusion at the involved level;
* Greater than grade 2 spondylolisthesis;
* Systemic infection or active infection at the surgical site;
* Active malignancy;
* Body Mass Index of 40 or higher;
* Significant metabolic bone disease (e.g. osteoporosis or osteomalacia) to a degree that spinal instrumentation is contraindicated;
* Taking medications that may interfere with bone or soft tissue healing (e.g. long-term steroid use);
* Alcohol or drug abuse;
* Waddell Signs of Inorganic Behavior >3;
* Currently in litigation regarding a spinal condition;
* Known sensitivity to implant material;
* A prisoner;
* Pregnant or contemplating pregnancy during the 24-month follow-up period; and
* Enrolled in another concurrent clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2003-07; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Krag, MD, Principal Investigator — Fletcher-Allen Health Center
Locations (11):
- United States (11):
  - Olympia Medical Center, Los Angeles, California
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - St. Mary's Christus Hospital, Shreveport, Louisiana
  - Providence Hospitals and Medical Center, Southfield, Michigan
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Alegent-Health Immanuel Medical Center, Omaha, Nebraska
  - St. Charles Hospital, Port Jefferson, New York
  - McLeod Health, Florence, South Carolina
  - Fletcher-Allen Health Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor — http://www.spineology.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Started | 123 | 33
Completed | 88 | 16
Not Completed | 35 | 17
Not completed — Lost to Follow-up | 35 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimesh 1500S | Structural Allograft Spacer | Total
Number analyzed (Participants) | 123 | 33 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 104 | 29 | 133
  >=65 years | 19 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.18 (12.19) | 53.91 (10.81) | 51.76 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 15 | 72
  Male | 66 | 18 | 84
Region of Enrollment [Number; unit: participants]
  United States | 123 | 33 | 156

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Low Back Pain Score at 24-months Compared to Pre-op
Description: A Visual Analog Scale (VAS) score was used to evaluate a subject's level of pain. The VAS is a 10 cm pain scale where a score of "0" represents "No Pain" and a score of "10" represents the "Worst Possible" pain. The magnitude of change in the 24-month score compared to the baseline score is calculated. A clinically meaningful change is defined as a 2 unit (cm) reduction at 24-months when compared to pre-op.
Time Frame: 24 month
Population: A total of 88 investigational and 16 control subjects completed this question at the 24-month timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 88 | 16
units on a scale | -4.0 (0.57825) | -4.0 (1.50207)

2. Primary Outcome: Mean Change in Back Function Score at 24-months Compared to Pre-op
Description: A subject's back function was assessed by the Oswestry Disability Index (ODI). The ODI is a 10 question survey that evaluates the degree of functional impairment. Completion of the survey yields a score from "0" to "100" points. A score of "0" represents "No disability" and "100" represents "Total disability". The magnitude of change between the two timepoints is reported. A clinically meaningful improvement is defined as a 15 point reduction at 24-months compared to the pre-op score.
Time Frame: 24 month
Population: A total of 88 investigational and 16 control subjects completed the ODI questionnaire at the 24-month timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 88 | 16
score on a scale | -21.6 (4.4055) | -18.4 (9.8028)

3. Primary Outcome: Number of Participants Determined to be a Fusion Success at 24 Months Post-operative
Description: Fusion Success is defined as <5 degrees angulation, <10% translation, and presence of bridging bone on CT.
Time Frame: 24 month
Population: A total of 77 investigational and 10 control subjects achieved the required imaging (x-rays and CT scan) at the 24-month timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 77 | 10
Participants | 71 | 10

4. Primary Outcome: Number of Participants With a Serious Device and Procedure Related Adverse Event
Description: The rate of serious device and procedure related adverse events are compared between the control and treatment arm from intraoperative through 24 months of follow-up.
Time Frame: From Intra-op through the 24-month visit
Measure: Count of Participants; unit: Participants
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 123 | 33
Participants | 14 | 6

5. Secondary Outcome: Right Leg Pain Score--Change From Preop at the 24-month Timepoint
Description: Right leg pain assessed by subject response on Visual Analog Scale (0-10 cm) where "0" represents "No pain" and "10" represents "Worst pain". The magnitude of change at 24-months compared to baseline is reported. A clinically relevant improvement is defined as a 2 cm reduction at 24-months compared to pre-op.
Time Frame: 24-month visit
Population: A total of 78 investigational subjects and 16 control subjects reported right leg pain scores at pre-op and 24-months postoperative.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 78 | 16
units on a scale | -2.6 (0.4) | -2.0 (0.6)

6. Secondary Outcome: Left Leg Pain--Change From Preop at the 24-month Timepoint
Description: Left leg pain assessed by subject response on Visual Analog Scale (0-10cm) where "0" represents "No left leg pain" and "10" represents "Worst Pain". The magnitude of change at 24-months post-operative compared to the baseline score is reported. A clinically relevant improvement is defined as a 2 cm reduction at 24-months compared to pre-op.
Time Frame: 24-month visit
Population: A total of 82 investigational subjects and 16 control subjects reported left leg pain scores at both pre-op and 24-months postoperative.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 82 | 16
units on a scale | -2.5 (0.4) | -2.5 (0.8)

7. Secondary Outcome: Number of Participants Rating Their Procedure as Very Satisfied or Somewhat Satisfied at 24-months Postoperative
Description: Subjects were asked to rate their satisfaction with their surgical procedure as "Very Satisfied", "Somewhat Satisfied", "Somewhat Dissatisfied" or "Very Dissatisfied" with their procedure
Time Frame: 24-month visit
Population: Patient satisfaction was not obtained in the early portion of this study. Therefore, a total of 39 investigational subjects and 16 control subjects that were enrolled in the latter portion of the study contributed responses to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
Number analyzed (Participants) | 39 | 16
Participants | 37 | 13

ADVERSE EVENTS:
Time Frame: Intraoperative through 24-months postoperative
Arm/Group | Optimesh 1500S | Structural Allograft Spacer
All-Cause Mortality (participants affected / at risk) | 3/123 | 0/33
Serious Adverse Events (participants affected / at risk) | 14/123 | 6/33
Other Adverse Events (participants affected / at risk) | 19/123 | 6/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Optimesh 1500S (N=123) | Structural Allograft Spacer (N=33)
Hematoma (Surgical and medical procedures) | 1 (1) | 0 (0) — Hematoma requiring evacuation
Pseudoarthrosis (Surgical and medical procedures) | 7 (9) | 1 (1)
Infection (Surgical and medical procedures) | 2 (2) | 1 (1) — Infection requiring Intervention
Adjacent Level Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Requiring Intervention
Screw Irritation (Surgical and medical procedures) | 3 (3) | 0 (0) — Requiring Intervention
Disc Herniation (Musculoskeletal and connective tissue disorders) | 2/2 (2) | 1 — Requiring Intervention
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Requiring Intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimesh 1500S (N=123) | Structural Allograft Spacer (N=33)
Lateral femoral cutaneous nerve injury secondary to intra-op positioning on table (Surgical and medical procedures) | 10 (10) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6)

LIMITATIONS AND CAVEATS:
1. This investigation was terminated early for protracted enrollment.
2. Multiple subjects were lost to follow-up at the 24-month visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No